CLINICAL TRIAL: NCT02941861
Title: Factors Influencing the 3-Year Recurrence of Liver Carcinoma After Surgery
Status: Completed | Type: Observational
Sponsor: Ruechuta Molek (Other)
Responsible Party: Sponsor-Investigator, Ruechuta Molek, Ms Ruechuta Molek (rmolek), Chulabhorn Hospital
Organization: Chulabhorn Hospital (Other)
Other Study IDs: 010/2016
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Liver Cancer; Recurrence
Keywords: Hepatocellular carcinoma; Cholangiocarcinoma; Recurrence
MeSH Terms: conditions — Liver Neoplasms; Recurrence; Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- recurrence rate of HCC after surgery: There were 33 for Hepatocellular carcinoma between February 2010 to December 2013. All patients were staged according to the tumor-node metastasis (TNM) system and appraised by the hospital tumor board conference. After surgery, an attending physician followed up patients by tumor marker and imaging as standard treatment as well as diagnosed its recurrence. In addition, all recurrence cases had standard treatments till the end of life. The survival was classified as the dates between the operation and the death.
  Interventions: Other: Recurrence Rate of HCC after surgery
- recurrence rate of CCA after surgery: There were 34 patients underwent liver resection for Cholangiocarcinoma between February 2010 to December 2013. All patients were staged according to the tumor-node metastasis (TNM) system and appraised by the hospital tumor board conference. After surgery, an attending physician followed up patients by tumor marker and imaging as standard treatment as well as diagnosed its recurrence. In addition, all recurrence cases had standard treatments till the end of life. The survival was classified as the dates between the operation and the death.
  Interventions: Other: Recurrence Rate of CCA after surgery

INTERVENTIONS:
Other: Recurrence Rate of HCC after surgery — Recurrence Rate of HCC after surgery
  Groups: recurrence rate of HCC after surgery
Other: Recurrence Rate of CCA after surgery — Recurrence Rate of CCA after surgery
  Groups: recurrence rate of CCA after surgery

SUMMARY:
Objective:

1. To study the factors that influence the 3- year recurrence of liver carcinoma after surgery
2. To study the related factors affecting recurrence of liver carcinoma after surgery

DETAILED DESCRIPTION:
Liver carcinoma including 80% Hepatocellular carcinoma (HCC) and 20% Cholangiocarcinoma (CCA) becomes the leading causes of death in East and South-East Asia. Though hepatectomy is the treatment of choice for early stage cancer, the recurrence has been reported as 30%, 62% and 79% in 1st, 3rd and 5th year respectively. Chulabhorn hospital, a cancer institute established in 2011, has been performing a 3-years retrospective study on the influencing factors and its correlation to liver carcinoma after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients underwent liver resection for Hepatiocellular carcinoma and Cholangiocarcinoma respectively including having pathology results between February 2010 to December 2013. Data was received from Cholabhron Hospital's patient database.

Exclusion Criteria:

* All patients having no pathology results were not included.
* All patients having no show for follow up recording were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There were 33 and 34 patients underwent liver resection for Hepatocellular carcinoma and Cholangiocarcinoma respectively between February 2010 to December 2013. All patients were staged according to the tumor-node metastasis (TNM) system and appraised by the hospital tumor board conference. After surgery, an attending physician followed up patients by tumor marker and imaging as standard treatment as well as diagnosed its recurrence. In addition, all recurrence cases had standard treatments till the end of life. The survival was classified as the dates between the operation and the death.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-08; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of Liver Carcinoma after surgery | 3 years

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Imamura H, Matsuyama Y, Tanaka E, Ohkubo T, Hasegawa K, Miyagawa S, Sugawara Y, Minagawa M, Takayama T, Kawasaki S, Makuuchi M. Risk factors contributing to early and late phase intrahepatic recurrence of hepatocellular carcinoma after hepatectomy. J Hepatol. 2003 Feb;38(2):200-7. doi: 10.1016/s0168-8278(02)00360-4. PMID 12547409
- [Background] Peduzzi P, Concato J, Kemper E, Holford TR, Feinstein AR. A simulation study of the number of events per variable in logistic regression analysis. J Clin Epidemiol. 1996 Dec;49(12):1373-9. doi: 10.1016/s0895-4356(96)00236-3. PMID 8970487
- [Background] Poon RT, Fan ST, Lo CM, Liu CL, Wong J. Intrahepatic recurrence after curative resection of hepatocellular carcinoma: long-term results of treatment and prognostic factors. Ann Surg. 1999 Feb;229(2):216-22. doi: 10.1097/00000658-199902000-00009. PMID 10024103
- [Background] Shimada M, Takenaka K, Taguchi K, Fujiwara Y, Gion T, Kajiyama K, Maeda T, Shirabe K, Yanaga K, Sugimachi K. Prognostic factors after repeat hepatectomy for recurrent hepatocellular carcinoma. Ann Surg. 1998 Jan;227(1):80-5. doi: 10.1097/00000658-199801000-00012. PMID 9445114
- [Background] Ko S, Nakajima Y, Kanehiro H, Hisanaga M, Aomatsu Y, Kin T, Yagura K, Ohyama T, Nishio K, Ohashi K, Sho M, Yamada T, Nakano H. Significant influence of accompanying chronic hepatitis status on recurrence of hepatocellular carcinoma after hepatectomy. Result of multivariate analysis. Ann Surg. 1996 Nov;224(5):591-5. doi: 10.1097/00000658-199611000-00001. PMID 8916872
- [Background] Hasegawa S, Ikai I, Fujii H, Hatano E, Shimahara Y. Surgical resection of hilar cholangiocarcinoma: analysis of survival and postoperative complications. World J Surg. 2007 Jun;31(6):1256-63. doi: 10.1007/s00268-007-9001-y. PMID 17453285
- [Background] Yusoff AR, Razak MM, Yoong BK, Vijeyasingam R, Siti ZM. Survival analysis of cholangiocarcinoma: a 10-year experience in Malaysia. World J Gastroenterol. 2012 Feb 7;18(5):458-65. doi: 10.3748/wjg.v18.i5.458. PMID 22346252
- [Background] Hanazaki K, Kajikawa S, Shimozawa N, Mihara M, Shimada K, Hiraguri M, Koide N, Adachi W, Amano J. Survival and recurrence after hepatic resection of 386 consecutive patients with hepatocellular carcinoma. J Am Coll Surg. 2000 Oct;191(4):381-8. doi: 10.1016/s1072-7515(00)00700-6. PMID 11030243
- [Background] Wadsworth CA, Dixon PH, Wong JH, Chapman MH, McKay SC, Sharif A, Spalding DR, Pereira SP, Thomas HC, Taylor-Robinson SD, Whittaker J, Williamson C, Khan SA. Genetic factors in the pathogenesis of cholangiocarcinoma. Dig Dis. 2011;29(1):93-7. doi: 10.1159/000324688. Epub 2011 Jun 17. PMID 21691113
- [Background] Portolani N, Coniglio A, Ghidoni S, Giovanelli M, Benetti A, Tiberio GA, Giulini SM. Early and late recurrence after liver resection for hepatocellular carcinoma: prognostic and therapeutic implications. Ann Surg. 2006 Feb;243(2):229-35. doi: 10.1097/01.sla.0000197706.21803.a1. PMID 16432356